CLINICAL TRIAL: NCT01827917
Title: Phase 4 Study of Speeda® Rabies Vaccinia That Use for Protection the Crowd Bitten by Animals to Three-level
Brief Title: The Protection Effect of Speeda® Rabies Vaccine for Human Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BJCDPC-6
Record Dates: First submitted 2013-03-27; First posted 2013-04-10 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2013-04

CONDITIONS: Rabies Vaccine Allergy
MeSH Terms: interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rabies vaccine (Experimental): When injured by the animal who carries the rabies virus, the patient after standard treatment would survive or die
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — Injection on day 0、7、21

SUMMARY:
The objective of this study was to achieve the post-marketing protective effect research of Speeda® rabies vaccine for human use from Chengda Bio.

DETAILED DESCRIPTION:
When found the injury who is bitten by the animal to three-level, the investigators would enroll the participant after explaining the protection and making him signed the informed consent. The patient would inject rabies vaccine as follow the national regulation, meanwhile the investigators would get the blood samples to detect whether the man-killer carries the rabies virus.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representatives of children or the adult participants are willing and able to understand the protocol requirements and provide informed consent signed
* Participant is considered to be in good health including the body and mental status on the basis of reported medical history and limited physical examination and live in local ≥ 12 months before injured
* The man-killer could found and detect whether it carries the virus

Exclusion Criteria:

* Known bleeding disorder or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Apply passive immunity preparation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Observation of the subject after injured by the animals carrying the virus | 2 years
  Whether or when would the patients develop symptoms after injured by the animals carrying the virus

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Principal Investigator — Beijing Chaoyang District Centers for Disease Control and Prevention
Locations (1):
- Hunan Centers for Disease Control and Prevention, Changsha, Hunan, China

REFERENCES:
- [Derived] Li L, Xu J, Zhang J, Wang F, Cai J, Yang L, Zhu Z, Bai Y, Jia B, Ma J, Shi N, Li S. Immunogenicity and immune persistence of Zagreb 2-1-1 regimen of rabies vaccine in Chinese healthy individuals: A randomized, parallel-controlled of homologous vaccine with different immune procedure study. Hum Vaccin Immunother. 2024 Dec 31;20(1):2403177. doi: 10.1080/21645515.2024.2403177. Epub 2024 Oct 2. PMID 39358206
- [Derived] Shi N, Zhang Y, Zheng H, Zhu Z, Wang D, Li S, Li Y, Yang L, Zhang J, Bai Y, Lu Q, Zhang Z, Luo F, Yu C, Li L. Immunogenicity, safety and antibody persistence of a purified vero cell cultured rabies vaccine (Speeda) administered by the Zagreb regimen or Essen regimen in post-exposure subjects. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-8. doi: 10.1080/21645515.2017.1279770. Epub 2017 Jan 25. PMID 28121231